CLINICAL TRIAL: NCT01630265
Title: Caregivers' Knowledge of Emergency Department Discharge Instructions Improves With the Use of Video
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Scott A. Bloch, Principal Investigator, Augusta University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 10-03-173
Record Dates: First submitted 2012-06-23; First posted 2012-06-28 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Evaluation of Video Discharge Instructions in Improving Understanding
Keywords: Discharge Instructions; Video Discharge Instructions; Video; Emergency Department Discharge Instructions; ED Discharge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Written Discharge Instructions (Active Comparator): Group of caregivers who read written discharge instructions that are the standard discharge instructions given in our pediatric ED
  Interventions: Other: Standard written discharge instructions
- Video Discharge Instructions (Experimental): Group of caregivers who watched the 3-minute video covering the information in the standard written discharge instructions
  Interventions: Other: Video Discharge Instructions

INTERVENTIONS:
Other: Standard written discharge instructions — Group of caregivers who read the standard written discharge instructions prior to answering the questionnaire
  Arms: Written Discharge Instructions
Other: Video Discharge Instructions — Group of caregivers who watched the 3 minute video covering the information in the standard written discharge instructions prior to answering the questionnaire
  Arms: Video Discharge Instructions

SUMMARY:
Previous studies demonstrate that patients often have difficulty understanding their discharge instructions. Video discharge instructions have the potential to mitigate factors such as illiteracy and limited physician time, which may affect comprehension. Our goal is to determine if adding video discharge instructions affects caregivers' understanding of their child's emergency department (ED) visit, plan and follow-up.

DETAILED DESCRIPTION:
Caregivers of patients, age 29 days to 18 years, with a diagnosis of fever, vomiting or diarrhea, and wheezing or asthma were randomized into written or video discharge instruction groups. In the ED, caregivers read standard written discharge instructions or watched a 3-minute video based on their child's diagnosis. They were then asked questions regarding information covered in these instructions. After completing the 20-point questionnaire, standard discharge procedure was followed. Caregivers were contacted by phone 2-5 days after discharge for a follow-up questionnaire. Usefulness of the discharge instructions was also assessed.

ELIGIBILITY:
Inclusion Criteria:

* caregivers of pediatric patients age 29 days to 18 years old diagnosed with wheezing or asthma exacerbation, fever, or vomiting and/or diarrhea.

Exclusion Criteria:

* Caregivers of patients who were critical in the ED,
* Admitted to the hospital, or given an alternate diagnosis prior to discharge were excluded from the study.
* Also, non-English speaking caregivers were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Knowledge about the child's diagnosis, treatment and follow-up care. | up to 5 days
  After reading standard written discharge instructions or watching a 3 minute video covering the information in the written discharge instructions, a questionnaire was completed by each caregiver. Knowledge was assessed based on the number of correct responses given by each caregiver at the time of ED discharge and 2-5 days post-discharge.

SECONDARY OUTCOMES:
Caregiver satisfaction with their discharge instructions | Satisfaction will be assessed at two time points within 5 days of being evaluated in the Emergency Department
  Caregivers either read standard written discharge instructions or watched a 3 minute video covering the information in the discharge instructions. Caregivers were then asked to rate their satisfaction with the discharge instructions using a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Bloch, MD, Principal Investigator — Augusta University
Locations (1):
- Medical College of Georgia, Augusta, Georgia, United States

REFERENCES:
- [Derived] Bloch SA, Bloch AJ. Using video discharge instructions as an adjunct to standard written instructions improved caregivers' understanding of their child's emergency department visit, plan, and follow-up: a randomized controlled trial. Pediatr Emerg Care. 2013 Jun;29(6):699-704. doi: 10.1097/PEC.0b013e3182955480. PMID 23714763